CLINICAL TRIAL: NCT02930512
Title: Study of Factors Associated With the Volumetric and Areal Bone Mineral Density and Bone Strength in Parkinson's Disease
Acronym: PAFOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0281; 2016-A00458-43 (Other: 2016-A00458-43)
Record Dates: First submitted 2016-10-07; First posted 2016-10-12 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Parkinson's Disease
Keywords: Bone mineral density; Osteoporosis; Parkinson's disease; Bone turnover markers
MeSH Terms: conditions — Parkinson Disease; Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- patients with idiopathic Parkinson's disease
  Interventions: Procedure: DXA scan; Procedure: pQCT scan

INTERVENTIONS:
Procedure: DXA scan
Procedure: pQCT scan

SUMMARY:
Studies show that patients with idiopathic Parkinson's disease (IPD) have an increased risk of fracture, particularly hip fracture whose complications and postoperative mortality appear to be higher than in the general population.

This increased risk of fracture is due partly to an increased risk of falling, and secondly to an impairment of bone tissue with lower bone mineral density (BMD). A meta-analysis concluded that patients with IPD have lower BMD than healthy controls. Prospective studies also showed rapid bone loss in these patients compared with controls. The association between low BMD and IPD seems dependent on the severity and duration of the disease even if some data are contradictory. Various mechanisms may explain this bone loss including weight loss, malnutrition and a low level of physical activity. However, enrollments in these studies are often weak and it is difficult to conclude on the real impact of these factors on bone loss in the IPD. The main objective of our study is to assess and prioritize from these various bone loss mechanisms. Bone assessment by "peripheral quantitative computed tomography" (pQCT) will also assess the impact of various risk factors on bone strength parameters. The prevalence of vertebral compression fractures in the IPD, at this day unknown can be evaluated. This study will also estimate the prevalence of vertebral compression fractures in the IPD.

DETAILED DESCRIPTION:
Studies show that patients with idiopathic Parkinson's disease (IPD) have an increased risk of fracture, particularly hip fracture whose complications and postoperative mortality appear to be higher than in the general population.

This increased risk of fracture is due partly to an increased risk of falling, and secondly to an impairment of bone tissue with lower bone mineral density (BMD). A meta-analysis concluded that patients with IPD have lower BMD than healthy controls. Prospective studies also showed rapid bone loss in these patients compared with controls. The association between low BMD and IPD seems dependent on the severity and duration of the disease even if some data are contradictory. Various mechanisms may explain this bone loss including weight loss, malnutrition and a low level of physical activity. However, enrollments in these studies are often weak and it is difficult to conclude on the real impact of these factors on bone loss in the IPD. The main objective of our study is to assess and prioritize from these various bone loss mechanisms. Bone assessment by "peripheral quantitative computed tomography" (pQCT) will also assess the impact of various risk factors on bone strength parameters. The prevalence of vertebral compression fractures in the IPD, at this day unknown can be evaluated. This study will also estimate the prevalence of vertebral compression fractures in the IPD.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic parkinson's disease (UKPDSBB criteria)
* Hoen and Yahr score < 4 (ON periods)
* Age between 35 and 70 years old
* Independent person at home

Exclusion Criteria:

* Dementia patient and progressive mental illness
* Patient with severe tremor
* Incapacity to walk over ten minutes
* Treatment influencing bone metabolism
* Disease influencing phosphocalcic metabolism
* Severe comorbidities
* Pregnant woman

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06-21 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Total bone mineral density of the tibia and radius quantified by peripheral quantitative computed tomography (pQCT) | at day 1

SECONDARY OUTCOMES:
Trabecular and cortical bone mineral density of the tibia and the radius | at day 1
Architectural parameters and bone resistance of the tibia and radius measured by pQCT | at day 1
Axial muscular area of the tibia and radius measured by pQCT | at day 1
Bone mineral density of the lumbar spine and hip measured by DXA | at day 1
body composition by DXA | at day 1
Parkinson's disease score | at day 1
Bone turnovers markers (CTX), 25 OH vitamin D | at day 1
Vertebral fracture assessment (VFA) | at day 1
Trabecular bone score of the lumbar spine | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine MALOCHET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France